CLINICAL TRIAL: NCT01967394
Title: Social Media, Teen Moms, and Postpartum Depression
Brief Title: Social Media, Teen Moms and PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mimia Logsdon, Professor, University of Louisville
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 1R15NR013563-01A1 (NIH); R15NR013563 (NIH)
Record Dates: First submitted 2013-10-10; First posted 2013-10-22 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Postpartum Depression
Keywords: Health Care Quality; Access; Evaluation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention County (Experimental): Use of internet based social marketing intervention
  Interventions: Other: Use of internet based social marketing intervention
- Control County (Placebo Comparator): No use of social media
  Interventions: Other: No use of social media

INTERVENTIONS:
Other: Use of internet based social marketing intervention — Eleven counties in Kentucky will be targeted with ads on Google and Facebook that direct adolescent mothers to an Internet-based social marketing intervention. The ads will be implemented using Facebook's and Google's ad network. The ads are setup, configured, and adjusted online. Facebook has identified key words that are recommended for adolescent mothers: "16 and pregnant," "teen mom,' and names of television shows with subject matter specific to adolescent mothers. We will target the ads to correspond to a geographical area that specifies a distance from the largest city in each county, and we will specify county lines. Ads will only appear on the Internet in the counties that are targeted for the intervention.
  Arms: Intervention County
Other: No use of social media — No social media ads will be available in these counties.
  Arms: Control County

SUMMARY:
Approximately 400,000 live births occur to adolescents in the United States annually. Of the 50% of adolescent mothers who experience depressive symptoms, less than 25% comply with referrals for depression evaluation and treatment due to lack of knowledge of depression symptoms (literacy), negative attitude towards mental health treatment, perception that individuals with depression are stigmatized (subjective norms), lack of understanding of health resources that are available to her and under her control (perceived control), and lack of time. Social media is a promising vehicle to reach and educate adolescent mothers since most adolescent mothers use social media for communication and to search for health information. Based upon the Theory of Planned Behavior, the investigators will target 11 counties in Kentucky with a social media ad campaign that will result in adolescent mothers (n=140) from those counties enrolling in an internet based intervention related to postpartum depression. The previously tested intervention includes vignettes from other adolescent mothers, questions and answers, resources, and an option to enroll in text message service. Before the intervention, after the intervention, and two weeks later the adolescent mothers will complete established questionnaires to determine if the intervention improved attitude and subjective norms towards depression and depression treatment, perceived control and intention related to seeking depression treatment, and the number of adolescent mothers with symptoms of depression who receive depression treatment. Data will be compared to scores on the same instruments from adolescent mothers (n=140) from the control group (18 other counties in Kentucky) that have not been targeted with the social media ad campaign or participated in the intervention. Data from the adolescent mothers in the control group will be collected in partnership with community agencies. The overall purpose of this trial is to test a cost effective and feasible method for reducing the cognitive and emotional barriers to accessing depression treatment in adolescent mothers. The specific aims are to (1) measure the extent to which a social media ad campaign is effective as a recruitment strategy; (2) test the effectiveness of an internet based social marketing intervention on both intention to seek treatment and rates of depression treatment, and (3) examine the dose effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Adolescent mothers, 13-21 years of age, who delivered a live child within the last 12 months, and has their baby residing with them. For the adolescent mothers enrolled in the Internet-based social marketing intervention, they must reside in Kentucky counties of Fayette, Jefferson, Bullitt, Henry, Oldham, Shelby, Spencer, Trimble, Christian, Warren or Barren. The adolescent mothers enrolled in the control group must reside in Kentucky counties of Campbell, Casey, Daviess, Boone, Nelson, Russell, Carroll, Kenton, Hardin, Hancock, Henderson, McClean, Meade, Ohio, Union, Webster, Meade or Marion

Exclusion Criteria:

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 287 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Social Marketing Intervention | 2 years
  How many teen mothers are enrolled in treatment programs for their depression per county? Is there a difference between counties?

SECONDARY OUTCOMES:
Number of teens seeking depression treatment | 2 years
  Do the teens in counties with the social media campaigns seek depression treatment more than those in the control counties.

OTHER OUTCOMES:
Intention of a adolescent to seek depression treatment | 2 years
  What is the association between intention to seek depression treatment and actual seeking of treatment, when controlling for baseline depression symptoms?

CONTACTS AND LOCATIONS:
Overall Officials: Mimia C Logsdon, PhD, Principal Investigator — University of Louisville
Locations (8):
- United States (8):
  - Three Rivers, Carrollton, Kentucky
  - Hands Program of Kenton County (Young Families of Children, Inc), Covington, Kentucky
  - Lincoln Trail Health Department, Elizabethtown, Kentucky
  - St. Joseph Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Hands Program of Boone and Campbell Counties (Every Child Succeeds), Newport, Kentucky
  - Three Rivers Health Department, Owensboro, Kentucky
  - Lake Cumberland Health Department, Somerset, Kentucky